CLINICAL TRIAL: NCT06149988
Title: A Phase I, Single Center Crossover Study, Evaluating the Pharmacokinetic Profile and Safety of Self-emulsified THC/CBD Powder Compared With Equivalent Dose of THC/CBD Oil, Orally Administered.
Brief Title: Comparative PK Study Of THC/CBD Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CapSoil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V1022022
Record Dates: First submitted 2023-10-22; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cannabis
Keywords: Powder; Oil
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose of THC/CBD S.E powder (Experimental): On visit 1: Subjects will receive a single dose of THC/CBD S.E powder- 500 mg, given orally.
  Interventions: Drug: THC/CBD S.E powder
- a single dose of THC/CBD oil (Active Comparator): On visit 2 (30 days later): Subjects will receive a single dose of THC/CBD oil- 8 mg, given orally (equivalent dose to the powder).
  Interventions: Drug: THC/CBD oil

INTERVENTIONS:
Drug: THC/CBD S.E powder — A single dose of THC/CBD S.E powder- 500 mg, given orally.
  Arms: Single dose of THC/CBD S.E powder
Drug: THC/CBD oil — Followed by a 30-day washout- A single dose of THC/CBD oil- 8 mg, given orally (equivalent dose to the powder).
  Arms: a single dose of THC/CBD oil

SUMMARY:
A phase I, single center crossover study.

The goal of this clinical trial is to learn about self-emulsified THC/CBD powder compared with equivalent dose of THC/CBD oil, orally administerd in healthy volunteers.

The main question it aims to answer is:

•If the pharmacokinetics profile of one dose of THC/CBD Self emulsified (S.E powder) compares to THC/CBD oil (equivalent dose).

The secondary is:

•If the use of THC/CBD S.E powder is tolerable and safe at least as THC/CBD oil.

Participants will receive a single dose of THC/CBD S.E powder followed by a 30-day washout period and then a single dose of THC/CBD oil.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 21-65 years old.
2. Subjects must have a signed study informed consent before any procedure.
3. Subjects must have a cannabis license as detailed at procedure No. 106 of the IMC-GCO , license will be issued and approved by PI at screening visit after signing on informed consent.
4. Female subjects must be of non-childbearing potential or, if of childbearing potential, must have a negative urine pregnancy test at screening, visit 1 and visit 2.

Exclusion Criteria:

1. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to THC/CBD.
2. Has an underlying medical condition that would preclude study participation.
3. Chronic use of medications for underlying medical conditions.
4. Use of any medications within 24 hours prior to treatment visit.
5. Is currently participating in another study of an investigational agent/medical device.
6. Has known psychiatric or substance abuse disorders that would interfere with participating in the study.
7. Patients who previously suffered from dysfunction of the: liver, kidneys, heart, blood vessels and immune system (such as transplant recipients or patients undergoing chemotherapy).
8. Patients who previously suffered from depression or anxiety.
9. Medical history of high blood pressure, low blood pressure or diabetes.
10. Patients who experience difficulties in performing daily activities.
11. Current cannabis use or positive THC urine test results.
12. Pregnant or lactating female subjects

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the pharmacokinetics profile of one dose of THC/CBD S.E powder compared to THC/CBD oil (equivalent dose): 1.a) THC/CBD S.E powder and oil exposure as measured by Cmax. | 30 days
  Measured by Cmax.
To demonstrate the pharmacokinetics profile of one dose of THC/CBD S.E powder compared to THC/CBD oil (equivalent dose): 1.b) THC/CBD S.E powder and oil exposure as measured by AUC. | 30 days
  Measured by AUC.
To demonstrate the pharmacokinetics profile of one dose of THC/CBD S.E powder compared to THC/CBD oil (equivalent dose): 2. THC/CBD S.E and oil powder half life | 30 days
  t1/2, should be determined by using model independent analytical methods.
To demonstrate the pharmacokinetics profile of one dose of THC/CBD S.E powder compared to THC/CBD oil (equivalent dose): 3. THC/CBD S.E powder and oil onset of action and time to reach maximum blood concentration as measured by Tmax. | 30 days
  Measured by Tmax.

SECONDARY OUTCOMES:
To demonstrate that the use of THC/CBD S.E powder is tolerable and safe at least as THC/CBD oil: Incidence of advert events (AEs), defined and graded according to the NCI-issued Common Terminology Criteria for Adverse Events (CTCAE). | though study completion, 30 days
  By tracking Incidence of advert events (AEs), defined and graded according to the NCI-issued Common Terminology Criteria for Adverse Events (CTCAE).

OTHER OUTCOMES:
Minimum blood concentration (Cmin) | though study completion, 30 days
  Cmin, by using model independent analytical methods.
Bioavailability | though study completion, 30 days
  By using model independent analytical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Vered Hermush, M.D., Principal Investigator — Laniado Hospital
Locations (1):
- Laniado Hospital, Netanya, Israel